CLINICAL TRIAL: NCT06429345
Title: Possible Role of Coenzyme Q10 in Prevention of Contrast Induced Nephropathy in Patients With Acute Coronary Syndrome Undergoing Coronary Angiography With or Without Intervention.
Brief Title: Coenzyme Q10 Role in Prevention of Contrast Induced Nephropathy in Acute Coronary Syndrome Patients.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS70/2024
Record Dates: First submitted 2024-03-19; First posted 2024-05-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Contrast-induced Nephropathy
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coenzyme Q10 100 Milligrams Oral Capsule (Experimental): Coenzyme Group received coenzyme Q10 in addition to the the standard preventive measures
  Interventions: Drug: Coenzyme Q10 100 Milligrams Oral Capsule
- Placebo group (Placebo Comparator): Placebo Group received only the standard preventive measures
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 100 Milligrams Oral Capsule — Patients will be randomly divided into two groups using a computer generated random number chart Coenzyme Q10 group will receive 400 milligrams coenzyme Q10 preoperative and 400 milligrams coenzyme Q10 for 3 days post operative in addition to the standard preventive measures.
  Other Names: Coenzyme Q10
  Arms: Coenzyme Q10 100 Milligrams Oral Capsule
Drug: Placebo — placebo group will receive only the standard preventive measures (as proper hydration pre and post operative)without the coenzyme Q10.
  Arms: Placebo group

SUMMARY:
In this study the investigators aim to study the effect of supplementation of CoQ10 in decreasing the incidence of contrast induced acute kidney injury in patients with acute coronary syndrome undergoing coronary angiography.

DETAILED DESCRIPTION:
Patients who fulfilled the inclusion criteria and agreed to participate in the study will be randomly divided into 2 groups using their computer generated random numbers that group a will receive the coenzyme Q10 in addition to the standard preventive measures and group b will receive only the standard preventive measures without the coenzyme Q10.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older.
* ST-elevation myocardial infarction (STEMI).
* Non ST-elevation myocardial infarction( NSTEMI).
* Unstable Angina (UA)

Exclusion Criteria:

* Renal transplant patients.
* Preoperative bleeding .
* Intraoperative bleeding or hypotension.
* Patients taking any nephrotoxic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of the Creatinine rise in 1st 48-72 hours in ccu | 48-72 hours
  a rise in serum creatinine of at least 0.5 mg/dL or a 25% increase from baseline within 48 to 72 hours after contrast exposure

CONTACTS AND LOCATIONS:
Overall Officials: RAMY Mohamed, Principal Investigator — Resident of cardiology department,Ain shams university
Locations (2):
- Egypt (2):
  - Ain Shams university hospitals, Cairo
  - Ramy Mohamed Mostafa, Cairo